CLINICAL TRIAL: NCT06009302
Title: Analgesic Effects of Extraoral Ultrasound Block of Mandibular Nerve for the Extraction of Lower Third Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Varazdin General Hospital (Other)
Collaborators: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12071987
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-08

CONDITIONS: Molar; Impacted Teeth
Keywords: dental anesthesia; inferior alveolar nerve; regional anesthesia; ultrasound; mandibular nerve
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US block of mandibular nerve (Experimental): Extraoral ultrasound-guided block of the mandibular nerve will be performed iusing an ultrasound device. After visualisation of the pterygomandibular space, of the maxillary artery and the mandibular nerve next to it, at a depth of 2-4 cm, the detection of the maxillary artery is confirmed by Color Doppler. A needle enters between the coronoid and condylar processes, using the "out of plane" technique, near the maxillary artery, and after negative aspiration, local anesthetic ropivacaine (0.75%, 2.5 mL) will be applied.
  Interventions: Procedure: US guided block of mandibular nerve
- intraoral block of lower alveolar nerve (Active Comparator): During the intraoral block of the inferior alveolar nerve, the patient will lie with his mouth wide open, and the inferior alveolar, lingual and buccal nerves will be anesthetized using two injections. The anesthetic used will be 40 mg/mL articaine chloride+0.01 mg/mL epinephrine: the planned amount of anesthetic is 2×1.7 mL, and if anesthesia is not achieved, an additional volume of anesthetic will be added as needed, until anesthesia
  Interventions: Procedure: Intraoral block of lower alveolar nerve

INTERVENTIONS:
Procedure: US guided block of mandibular nerve — Extraoral ultrasound-guided block of the mandibular nerve will be performed in the examined group using an ultrasound device, using ropivacaine (0.75%, 2.5 mL).
  Arms: US block of mandibular nerve
Procedure: Intraoral block of lower alveolar nerve — Block of lower alveolar nerve will be applied intraoraly using articaine+adrenaline
  Arms: intraoral block of lower alveolar nerve

SUMMARY:
This is a study about the dynamics and effects of different types of blocks (intraoral conduction anesthesia of the alveolar nerve and extraoral US block of the mandibular nerve) for extraction of lower third molars.

DETAILED DESCRIPTION:
Standard method of anesthesia for extraction of horizontally positioned lower thirdmolars is intraoral conduction anesthesia of the inferior alveolar nerve. However, the analgesiceffect of block is short and it is necessary to use analgesics. In this prospective clinical study,analgesic effect of ultrasound (US) -guided extraoral block of mandibular nerve will beinvestigated, in order to prolong pain-free time and reduce the use of analgesics associated withrisks (bleeding, hepatotoxicity).

Characteristics of alveolar nerve block and US block of the mandibular nerve will becompared, such as: pain during application of anesthesia, amount of anesthetic, duration ofanesthesia, need to use analgesics, time to and level of pain when using analgesics, andcomplications

ELIGIBILITY:
Inclusion Criteria:

* age 18-64 years
* horizontally placed lower third molars
* ASA I or II group

Exclusion Criteria:

* allergy to local anesthetics
* local infection at the site of needle puncture
* parotitis
* serious liver disease
* use of antiarrhythmics group III (eg amiodarone), anticoagulant or antithrombotic drugs
* lactation
* people who took an analgesic as a preventive measure before coming to the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Time without pain | first 24 postoperative hours

SECONDARY OUTCOMES:
Time of numbness | first 24 postoperative hours
Pain level when anesthesia is applied | first 24 postoperative hours
  0-10 on VAS
Pain level when painkiller is needed | first 24 postoperative hours
  0-10 on VAS

CONTACTS AND LOCATIONS:
Locations (1):
- Varazdin General Hospital, Varaždin, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khorshidi Khiavi R, Pourallahverdi M, Pourallahverdi A, Ghorani Khiavi S, Ghertasi Oskouei S, Mokhtari H. Pain control following impacted third molar surgery with bupivacaine irrigation of tooth socket: a prospective study. J Dent Res Dent Clin Dent Prospects. 2010 Fall;4(4):105-9. doi: 10.5681/joddd.2010.027. Epub 2010 Dec 21. PMID 23346335
- [Background] Fisher SE, Frame JW, Rout PG, McEntegart DJ. Factors affecting the onset and severity of pain following the surgical removal of unilateral impacted mandibular third molar teeth. Br Dent J. 1988 Jun 11;164(11):351-4. doi: 10.1038/sj.bdj.4806453. No abstract available. PMID 3165011
- [Background] Teoh L, Moses G, McCullough MJ. A review of drugs that contribute to bleeding risk in general dental practice. Aust Dent J. 2020 Jun;65(2):118-130. doi: 10.1111/adj.12751. Epub 2020 Mar 13. PMID 32064612
- [Background] Plantevin F, Pascal J, Morel J, Roussier M, Charier D, Prades JM, Auboyer C, Molliex S. Effect of mandibular nerve block on postoperative analgesia in patients undergoing oropharyngeal carcinoma surgery under general anaesthesia. Br J Anaesth. 2007 Nov;99(5):708-12. doi: 10.1093/bja/aem242. Epub 2007 Sep 19. PMID 17884802
- [Background] Kumar A, Sinha C, Kumar A, Kumari P, Mukul SK. Ultrasound-guided trigeminal nerve block and its comparison with conventional analgesics in patients undergoing faciomaxillary surgery: Randomised control trial. Indian J Anaesth. 2018 Nov;62(11):871-875. doi: 10.4103/ija.IJA_256_18. PMID 30532323
- [Background] Stojanovic S, Buric N, Tijanic M, Todorovic K, Buric K, Buric N, Jovanovic M, Bajagic V. The Assessment of Prolonged Inferior Alveolar Nerve Blockade for Postoperative Analgesia in Mandibular Third Molar Surgery by a Perineural Addition of Dexamethasone to 0.5% Ropivacaine: A Randomized Comparison Study. Int J Environ Res Public Health. 2022 Jan 25;19(3):1324. doi: 10.3390/ijerph19031324. PMID 35162346
- [Derived] Martinus M, Mihaljevic S, Reiner K, Verzak Z, Panic MK, Strahija A, Gluncic V, Lukic IK, Lukic A. Analgesic effect of ultrasound-guided extraoral mandibular nerve block compared to intraoral conductive block of the inferior alveolar nerve after lower third molar alveolectomy: a clinical prospective study. BMC Oral Health. 2024 Sep 4;24(1):1041. doi: 10.1186/s12903-024-04787-5. PMID 39232703
- See also: Side effect of glucosaimine to coagulation — https://halmed.hr/upl/lijekovi/PIL/Arthryl-1500-mg-prasak-za-oralnu-otopinu-PIL.pdf
- See also: The use of analgesics and anti-inflammatories in an oral surgery service in Medellín, Colombia, 2013-2015 — http://www.scielo.org.co/scielo.php?script=sci_arttext&pid=S0121-246X2019000100166